CLINICAL TRIAL: NCT03162328
Title: A Double-Blind Placebo-Controlled Multi-Site Randomized Cross-Over Study of the Effectiveness and Efficacy of the PowerSleep Device
Brief Title: A Study of the Effectiveness and Efficacy of the PowerSleep Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AI-16128-PSPIV-LO
Record Dates: First submitted 2017-05-16; First posted 2017-05-22 (Actual); Results first posted 2019-01-29 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Sleep Deprivation; Insufficient Sleep Syndrome; Healthy
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled cross-over study
Who Masked: Participant, Investigator
Masking Description: Participants are randomized to two different therapies: Sham or Stimulation. Sites are masked as they are randomized to: Therapy A or Therapy B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Powersleep Sham, PowerSleep Stim (Placebo Comparator): Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers. After 2 nights in the lab in the sham condition participants will cross-over to the other arm of the trial the following week. Week 2 - Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night.
  Interventions: Device: PowerSleep Stim; Device: PowerSleep Sham
- Powersleep Stim, PowerSleep Sham (Experimental): Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night. After 2 nights in the lab in the stim condition participants will cross-over to the other arm of the trial the following week. Week 2 - Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers.
  Interventions: Device: PowerSleep Stim; Device: PowerSleep Sham

INTERVENTIONS:
Device: PowerSleep Stim — Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night.
Device: PowerSleep Sham — Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers.

SUMMARY:
This study is a randomized, double-blind, placebo-controlled cross-over study designed to evaluate the effectiveness and efficacy of 2 consecutive work days of nightly use of active versus sham PowerSleep devices in adults with self-imposed restricted sleep schedules. The primary analysis will be intent-to-treat with the secondary analysis as an as-treated analysis. The expected duration of the study for each participant is up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to admission
* Able to read, write and speak English
* Adult volunteers aged 21-50 years
* Working full time with a regular work schedule; Full time is considered 4- 10 hour days or 5- 8 hour days with a start time of 7am or later
* Self-reported regular sleep schedule who are able to maintain their sleep schedule during the course of the study
* Self-reported sleep duration of > 5hrs. and ≤ 7 hrs. +/- 15 minutes (verified by 6 work days of ambulatory sleep monitoring with wrist actigraphy and daily logs)
* Self-reported sleep latency > 30 minutes no more than once / wk. (time to fall asleep)
* Self-reported wake time after sleep onset ≤ 30 minutes
* Participants who regularly use an alarm clock during the work week and who self-report:

  i. Regular time in bed (TIB) on work days of ≤7 hours ii. Regular increase in sleep duration by ≥ 1 hour during non-work days as compared to work days, either by nocturnal bedtime extension of via a daytime nap

Exclusion Criteria:

* Participation in another interventional study in the past 30 days.
* Previously enrolled in a PowerSleep study.
* Major controlled* or uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure, cancer, Chronic Obstructive Pulmonary Disease (COPD), respiratory failure or insufficiency, or patients requiring oxygen therapy (as determined by self-report and reviewed by the study PI.)
* Currently working night, swing, split or rotating shift.
* Current use or use of within the past month of a prescription or over-the-counter sleep medication or stimulant; use of psychoactive medication (based on self-report and review with a study clinician). Refer to table below for examples.
* Pregnant or currently breast feeding
* Current Smokers or using nicotine replacement therapy. Those that have been nicotine free for 30 days will be included.
* Body Mass Index > 40 kg/m2
* Prior diagnosis of any sleep disorder including

  1. Obstructive Sleep Apnea (AHI ≥15 events/hour) - from ambulatory or in lab polysomnography
  2. Restless legs syndrome, or periodic limb movement disorder
  3. Insomnia
  4. Parasomnia
* High Risk of Obstructive Sleep Apnea (OSA) based on STOP-BANG Questionnaire ("yes" on at least 4 of 8 questions)
* High Risk of Restless Legs Syndrome (RLS) based on Cambridge-Hopkins Screening questionnaire
* High Risk of Insomnia based on Insomnia Severity Index (score of 22 or higher)
* Self-reported history of excessive alcohol intake- self-report > 21 drinks / wk or binge alcohol consumption ( >5 drinks per day)
* Excessive caffeine consumption (> 650mg/day combining all caffeinated drinks regularly absorbed during workdays.) Caffeine intake must be regular and maintained throughout study and on testing days
* Individuals who self-report a history of recurrent seizures or epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion).
* Individuals who self-report severe contact dermatitis or allergy to silicone, nickel or silver.
* Individuals who self-report moderate hearing loss.
* Inability to achieve appropriate headband fit.
* Planned travel across more than one time zone one month prior to and or during the anticipated period of the study with PowerSleep device use
* Intentional naps during the work week.
* Alpha-Delta waveforms as determined by Baseline night PowerSleep Device data collection

  * Participants who are on a stable and well-tolerated pharmacological treatment for hypertension, dyslipidemia, or thyroid replacement will not be excluded as long as they continue to take their medication at the same dose and at the same time(s) of day.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Arkansas Center for Sleep Medicine, Little Rock, Arkansas
  - Florida Lung & Sleep Associates, Lehigh Acres, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Clayton Sleep Institute, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No, this data will remain within Philips Respironics.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 participants across 7 sites were screened for eligibility for this study. Recruitment was open April 2017 through November 2017.
Pre-assignment Details: Of the 84 participants screened, 63 were found to be eligible,however 1 eligible participant withdrew at the randomization visit, but prior to randomization. 1 participant withdrew after being randomized. 1 participant did not complete all study visits, but had enough device data to be included in the analysis.
Groups:
- Screening Population: All patients that signed consent are considered for the screening population.
Period: Screening Period
Arm/Group | Screening Population | Powersleep Sham, PowerSleep Stim | Powersleep Stim, PowerSleep Sham
Started | 84 | 0 | 0
Completed | 62 | 0 | 0
Not Completed | 22 | 0 | 0
Not completed — Did not meet inclusion/exclusion | 21 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Study Period
Arm/Group | Screening Population | Powersleep Sham, PowerSleep Stim | Powersleep Stim, PowerSleep Sham
Started | 0 | 30 | 32
Completed | 0 | 30 | 31
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients that were consented where consented for this study are considered for the screening population.
Arm/Group | Screening Population
Number analyzed (Participants) | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 84
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.70 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 55
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 84
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.79 (5.14)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 71.38 (10.77)
Blood Pressure- Systolic [Mean (Standard Deviation); unit: mmHg] | 118.80 (15.71)
Blood Pressure- Diastolic [Mean (Standard Deviation); unit: mmHg] | 76.42 (10.58)
Epworth Sleepiness Scale Total [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale is an 8 item questionnaire that measures the general level of daytime sleepiness. Participants were asked what the chance is they would doze off or fall asleep during different routine daytime situations. The survey answers questions on a scale of 0 to 3- 0 being no chance and 3 being a high chance of dozing. The lowest score possible is a 0 and the highest score possible is a 24.
  units on a scale | 5.48 (3.74)
insomnia severity index [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) has seven questions about sleep problems. The answers are scored 0 to 4 and added to obtain a total score which indicates the clinical significance of the insomnia complaint. Total score can range from 0 (no clinically significant) to 28 (clinical insomnia, severe).
  units on a scale | 7.31 (5.33)
Temperature [Mean (Standard Deviation); unit: degrees Farenheit] | 97.76 (0.89)
Weight [Mean (Standard Deviation); unit: pounds] | 172.48 (41.80)
Neck Circumference [Mean (Standard Deviation); unit: centimeters] | 35.09 (3.93)

OUTCOME MEASURES:

1. Primary Outcome: Average Amount of Slow Wave Activity Delivered by the Powersleep Device With and Without Stimulation
Description: It is hypothesized that the use of active PowerSleep over two work nights of use, as compared to the sham device over two work nights of use, will result in a significant increase (≥5%), in mean total slow-wave activity (SWA). Slow wave activity (SWA) corresponds to the EEG power in the 0.5 to 4 Hz band during non-rapid eye movement (NREM) sleep. SWA reflects the number and amplitude of slow-waves and determines the speed with which sleep-need dissipates.
Time Frame: 4 nights
Population: 5 data sets were lost in the Sham/Stim condition: 1 - noisy data, 4 - not crossed over 4 data sets were lost in the Stim/Sham condition: 4 - not crossed over
Measure: Mean (Standard Deviation); unit: microvolts^2
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 52 | 52
microvolts^2 | 1649.41 (896.05) | 1643.84 (847.34)
Statistical Analysis 1: Comparison: Powersleep Sham vs PowerSleep Stim; Test type: Superiority; p = 0.363, Wilcoxon Signed Ranks Test

2. Primary Outcome: Cumulative Amount of Slow Wave Activity Delivered by the Powersleep Device With and Without Stimulation
Description: It is hypothesized that the use of active PowerSleep over two work nights of use, as compared to the sham device over two works nights of use, will result in a significant increase (≥5%), in mean total slow-wave activity (SWA).The integral of SWA (CSWA) over a sleep session, is directly proportional to the sleep-need dissipation occurring during said sleep session.
  In our research, both SWA and CSWA are evaluated as relative values having as reference the average SWA and CSWA over sham sleep sessions. CSWA is the integral of SWA which is why the unit of CSWA is microvolt^2×minute.
Time Frame: 4 nights
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microvolts^2×minute
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 52 | 52
microvolts^2×minute | 1437304 (1290198) | 1444740 (1220632)
Statistical Analysis 1: Comparison: Powersleep Sham vs PowerSleep Stim; Test type: Superiority; p = 0.291, Wilcoxon Signed Ranks Test

3. Secondary Outcome: Changes in Multiple Sleep Latency Test (MSLT)
Description: To evaluate the relationship between MSLT (sleep latency) and changes in SWA. This evaluated the average length of time it took a participant to fall asleep (in minutes) for each of the 4 naps in each condition, after two nights of sham and two nights of stim.
Time Frame: 4 nights
Population: 1 participant was excluded from the analysis because of a nap in between treatment nights
  1 participant was excluded from the analysis because they did not complete the final night of the study 4 data sets were lost in the Sham/Stim condition: 4 - not crossed over 4 data sets were lost in the Stim/Sham condition: 4 - not crossed over
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 51 | 51
minutes | 10.3 (5.4) | 10.3 (5.3)

4. Secondary Outcome: Paired Associates Learning (PAL)
Description: To measure trends of memory of 2 weeks of home use randomized with active PowerSleep (delivering audio tones) as compared to a two weeks of sham (delivering no audio tones).
  Participants answered completed an 80 word pair memory recall in the morning following the overnight in the sleep lab. The results listed below are the mean and standard deviation of the PowerSleep treatment week compared to the Sham treatment week. Learning was completed on the last night in the lab in each arm, with recall in the morning.
  PAL Differences (morning - evening responses): Difference between number correct the morning recall and the evening recall
  Correct Responses (evening recall): number of correct responses during the evening recall
  Correct Responses (morning call): number of correct responses during the morning recall, after the night in the sleep lab.
Time Frame: 4 nights
Population: 1 participant was excluded from the analysis because they did not complete the final night of the study 4 data sets were lost in the Sham/Stim condition: 4 - not crossed over 4 data sets were lost in the Stim/Sham condition: 4 - not crossed over
  1 participant did not complete the learning in the evening therefore data was unscorable.
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | Powersleep Sham | Powersleep Stim
Number analyzed (Participants) | 51 | 51
number of words
  PAL Differences (morning - evening responses) | 7.45 (8.38) | 8.51 (7.5)
  Correct Responses (evening recall) | 21.76 (10.74) | 23.82 (14.37)
  Correct Responses (morning recall) | 29.22 (12.11) | 32.33 (17.19)

5. Secondary Outcome: Changes in Cognitive Testing - Verbal Fluency
Description: To evaluate the relationship between cognitive testing changes and changes in SWA. Verbal fluency is a type of cognitive testing in which participants are required to generate as many words directly related to the instructions as they can. This task has three conditions each arm:letter fluency (F,A,S and B,H,R),category fluency (Animals, Boys names and clothing girls names) and category switching (Fruits and furniture and vegetables and musical instruments). Each trial with each condition lasts for 60 seconds.
  Total correct responses are calculated by counting the number of correct words generated for each condition: letter fluency, category fluency and switching
  Total repetition errors are calculated by counting any response that is repeated within the 60sec trial for each condition.
  Total set-loss errors are any response that violates any of the criterion rules of the condition (for example saying Bill instead of Beth for girls names) for each condition.
Time Frame: 4 nights
Population: 5 participants did not have verbal fluency recorded therefore were unable to be scored
  1 participant was excluded from the analysis because they did not complete the final night of the study
  1 participant was excluded because they had to repeat second work week 8 data sets were lost because they were not crossed over
Measure: Mean (Standard Deviation); unit: words
Groups:
- Powersleep Stim: Participants will wear the PowerSleep device with soft audio tones administered via the speakers during deep sleep throughout the night. After 2 nights in the lab in the stim condition participants will cross-over to the other arm of the trial the following week. Week 2 - Participants wear the same PowerSleep device as with the active treatment, however no audio tones will be administered via the speakers.
Arm/Group | Powersleep Sham | Powersleep Stim
Number analyzed (Participants) | 46 | 46
words
  Category Fluency - Total Correct | 42.5 (8.15) | 42.52 (7.77)
  Category Fluency - Total Repetition Errors | 1.04 (1.11) | 0.74 (1.06)
  Category Fluency - Total Set Loss Errors | 0.7 (1.59) | 0.61 (1.16)
  Category Switching - Number Correct | 14.67 (2.25) | 13.8 (2.55)
  Category Switching - Number of Repetition Errors | 0.17 (0.49) | 0.39 (0.71)
  Category Switching - Number of Set Loss Errors | 0.35 (0.74) | 0.37 (0.80)
  Letter Fluency - Total Correct | 38.28 (9.36) | 38.72 (11.35)
  Letter Fluency - Total Repetition Errors | 0.98 (1.29) | 1.26 (1.5)
  Letter Fluency - Total Set Loss Errors | 0.63 (0.9) | 0.41 (1.15)

6. Secondary Outcome: Average Subjective Sleepiness Scales.
Description: Average subjective sleepiness scales, as measured by scores on a scale of 0 to 10, PowerSleep Sham over 2 works nights of use as compared to PowerSleep Stim over 2 works nights of use. For these outcomes the 0 was the worst, 10 being the best.
  Sleepiness scales were completed each morning following after the 2 nights of the one condition and the 2 nights in the other condition. The values of 2 nights (mornings after) are averaged and compared to the average of the 2 nights the following week. Therefore the timeframe is 4 nights.
Time Frame: 2 days following each intervention, over 9 days
Population: 8 data sets were lost in the analysis as participants were randomized but not crossed over to the other arm of the study.
  1 data set was lost because the wrong form was administered.
  1 participant did not complete the final overnight
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 51 | 51
score on a scale
  How alert you feel? | 6.36 (2.18) | 6.61 (2.19)
  How deep was your sleep? | 6.25 (2.13) | 6.52 (1.99)
  How mentally refreshed you feel? | 6.35 (2.07) | 6.68 (2.11)
  Rate your sleep quality? | 6.18 (2.11) | 6.38 (2.08)

7. Secondary Outcome: Average Subjective Sleepiness Scale- Karolinska Sleepiness Scale
Description: Average subjective sleepiness between PowerSleep Sham nights as compared to PowerSleep Stim nights on the Karolinska Sleepiness Scale 1 - very alert, 9 - very sleepy, great effort to keep awake
  Sleepiness scales were completed each morning following after the 2 nights of the one condition and the 2 nights in the other condition. The averages of the 2 nights (mornings after) are compared to the averages of the 2 nights (mornings after) the following week. Therefore the timeframe is 4 nights.
Time Frame: 2 days following each intervention, over 9 days
Population: 4 data sets were lost in the Sham/Stim condition: 4 - not crossed over 4 data sets were lost in the Stim/Sham condition: 4 - not crossed over
  1 participant napped between overnights and was excluded from the daytime measures
  1 participant did not complete the final overnight
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 51 | 51
score on a scale | 3.97 (1.62) | 3.76 (1.97)

8. Secondary Outcome: Average of Subjective Sleepiness Scale- Samn Perelli
Description: Average subjective sleepiness between PowerSleep Sham as compared to PowerSleep Stim on the Samn Perelli questionnaire 1 - fully alert, wide awake, extremely peppy and 7 - completely exhausted, unable to function effectively, ready to drop
  Sleepiness scales were completed each morning following after the 2 nights of the one condition and the 2 nights in the other condition. The averages of the 2 nights (mornings after) are compared to the average of the 2 nights(mornings after) the following week. Therefore the timeframe is 4 nights.
Time Frame: 2 days following each intervention, over 9 days
Population: 8 data sets were lost as participants were not crossed over to the other arm of the trial.
  1 participant napped between overnights and was excluded from the daytime measures
  1 participant did not complete the final overnight
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 51 | 51
score on a scale | 3.07 (1.06) | 2.88 (1.26)

9. Secondary Outcome: Psychomotor Vigilance Test - Reaction Times
Description: To measure trends of vigilance of (2 nights) of home use randomized with active PowerSleep (delivering audio tones) as compared to (2 nights) of sham (delivering no audio tones). This measured how quickly participants reacted to visual stimulus.
  Reaction time is the latency at which the participant reacts to a visual stimulus > 100 ms.
Time Frame: 4 nights
Population: 2 participants completed the wrong PVT
  1 participant did not complete the final overnight
  1 participant did not complete the PVT after wake-up 8 data sets were lost as participants did not cross over
  1 participant napped in between overnights and the data was no usable
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Powersleep Sham: All participants who wore the PowerSleep deice in the sham condition for at least one night.
- PowerSleep Stim: All Participants who wore the PowerSleep device in the Stim condition.
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 48 | 48
milliseconds
  Average 10% fastest reaction time | 192.59 (14.68) | 187.97 (16.72)
  Average reaction time | 258.77 (32.78) | 254.24 (38.00)
  Average 10% slowest reaction time | 433.16 (128.13) | 428.07 (180.61)

10. Secondary Outcome: Psychomotor Vigilance Test - Number of Anticipation and Number of Lapses.
Description: To measure trends of vigilance of (2 nights) of home use randomized with active PowerSleep (delivering audio tones) as compared to (2 nights) of sham (delivering no audio tones). Anticipations are the increase in errors of commission (responses without a stimulus) response time <100ms. Lapses (errors of omission) are measured or usually defined as reaction Times ≥ 500 ms.
Time Frame: 4 nights
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: count of events
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 48 | 48
count of events
  Number of anticipations | 4.35 (5.29) | 5.77 (10.92)
  Number of Lapses | 4.9 (5.2) | 3.9 (4.83)

11. Secondary Outcome: Psychomotor Vigilance Test - Average Speed
Description: To measure trends of vigilance of (2 nights) of home use randomized with active PowerSleep (delivering audio tones) as compared to (2 nights) of sham (delivering no audio tones). This measured the average speed with which participants respond to a visual stimulus. The average speed is 1/RT (also called reciprocal response time or response speed).
Time Frame: 4 nights
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: 1/s
Arm/Group | Powersleep Sham | PowerSleep Stim
Number analyzed (Participants) | 48 | 48
1/s | 4.14 (0.43) | 4.22 (0.39)

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected over a 6 week period
Description: An adverse event (AE) is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study device, whether or not considered related to study device.
  AEs will include:
  * Changes in the general condition of the participant
  * Subjective symptoms offered by or elicited from the participant;
  * Signs observed by the investigator or study personnel;
Groups:
- Screening Period: All Study participants that were consented to the study.
Arm/Group | Screening Period | PowerSleep Sham, PowerSleep Stim | Powersleep Stim, PowerSleep Sham
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 0/84 | 0/30 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03162328/Prot_SAP_000.pdf